CLINICAL TRIAL: NCT06571552
Title: Description of Coagulation Disorders Secondary to Two Plasmapheresis Techniques (Double Filtration Plasmapheresis vs. PFS). Descriptive Pilot Study.
Brief Title: Coagulation Disorders Secondary to Two Plasmapheresis Techniques (Double Filtration Plasmapheresis vs. PFS). Descriptive Pilot Study.
Acronym: APHERCOAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: NIMAO/2023-2/OM01
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hyperfibrinogenemia; Hemostatic Disorder
Keywords: Double Filtration Plasmapheresis; Single Plasma Exchange
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Patients being monitored for chronic therapeutic plasmapheresis with regional citrate anticoagulation will be recruited from the Nephrology Department at Nîmes University Hospital. After receiving written informed consent (inclusion visit), patients will be randomized to determine the nature of their first cycle (single plasma exchange or double filtration plasmapheresis. The next cycle will vary accordingly: DFPP if the first cycle was single plasma exchange, and single plasma exchange if the first session was DFPP.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients benefitting from Single Plasma Exchange followed by Double Filtration Plasmapheresis (Active Comparator): For the patients in this group, the first cycle (T1) will consist of Single Plasma Exchange and the second cycle (T2) of Double Filtration Plasmapheresis.
  Interventions: Procedure: Single Plasma Exchange followed by Double Filtration Plasmapheresis
- Patients benefitting from Double Filtration Plasmapheresis followed by Single Plasma Exchange (Active Comparator): For the patients in this group, the first cycle (T1) will consist of Double Filtration Plasmapheresis and the second cycle (T2) of Single Plasma Exchange.
  Interventions: Procedure: Single Plasma Exchange followed by Double Filtration Plasmapheresis

INTERVENTIONS:
Procedure: Single Plasma Exchange followed by Double Filtration Plasmapheresis — Double Filtration Plasmapheresis followed by Single Plasma Exchange

SUMMARY:
Therapeutic plasmapheresis causes changes in haemostasis by purifying many of the circulating factors involved. Few reliable data are available on these changes and most studies are limited to coagulation factor assays before and after the session, with little data documenting the kinetics of regeneration of these factors. It is recognized that haemostasis disorders caused by therapeutic apheresis must be corrected in cases of active bleeding. However the methods of correcting these disorders are debatable. Finally, it is unclear when changes in haemostasis associated with coagulation factor deficiency should be corrected. Haemostasis is probably not based solely on the level of blood fibrinogen, but it is most often its threshold that is used to trigger replacement therapy to prevent a supposed risk of haemorrhage. No studies are available on the kinetics of haemostasis disorders and the risk of haemorrhage following a therapeutic plasmapheresis session, according to session type and fibrinogen level at the end of the session. The hypothesis of this research is that the link between fibrinogen level and thrombin generation capacity, post therapeutic plasmapheresis, will enable us to better assess the risk of haemorrhage and propose preventive measures.

DETAILED DESCRIPTION:
Therapeutic plasmapheresis causes changes in haemostasis by purifying many of the circulating factors involved. Some data are available on changes in circulating haemostasis factors with the Single Plasma Exchange technique and the Double Filtration Plasmapheresis; however, most often these studies are carried out in specific clinical situations where other haemostasis disorders may be present, such as severe renal failure. Furthermore, in these studies, assessment of changes in haemostasis is often limited to coagulation factor assays before and after the session, with little data documenting the kinetics of regeneration of these factors, whose molecular weight and half-life vary widely. To date, there is no clear consensus/recommendation on the management of haemostasis disorders secondary to therapeutic apheresis. The need to correct haemostasis disorders caused by therapeutic apheresis also appears to be consensual in cases of active bleeding.The methods of correcting haemostasis disorders can also be discussed between infusion of coagulation factor and fresh frozen plasma. Finally, apart from these clinical situations, it is not clear when changes in haemostasis associated with coagulation factor deficiency should be corrected. There are no studies available on the kinetics of haemostasis disorders and the risk of haemorrhage following a therapeutic plasmapheresis session, depending on the type of session and the fibrinogen level at the end of the session. The hypothesis of our research is that the existence of a link between fibrinogen level and thrombin generation capacity, post therapeutic plasmapheresis, will enable us to better assess the risk of haemorrhage and to propose preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients without renal failure treated with chronic therapeutic plasmapheresis with a minimum treatment interval of 10 days and who can be treated with single plasma exchange (SPE) or double filtration plasmapheresis (DFPP) in accordance with the international recommendations.
* Therapeutic plasmapheresis with regional citrate anticoagulation.
* Patients over 18 years of age.
* Patient affiliated to or benefiting from a social security scheme.
* Free, informed and written consent, signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patients treated with oral anticoagulants or anti-platelet agents.
* Patients treated for hypercholesterolaemia or hypertriglyceridaemia; hyperviscosity, acquired haemophilia or nephrotic syndrome.
* Indication for substitution with fresh frozen plasma (FFP) for the treatment of the disease.
* Patient in an exclusion period determined by another study.
* Patient under court protection, guardianship or curatorship.
* Patient unable to give consent.
* Patient for whom it is impossible to give informed information.
* Pregnant or breast-feeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Determination of fibrinogen levels before the first plasmapheresis session with single plasma exchange | Day 0, before the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® before the first plasmapheresis session with single plasma exchange | Day 0, before the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the first plasmapheresis session with single plasma exchange | Day 0, end of session
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® after the first plasmapheresis session with single plasma exchange | Day 0, end of session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the plasmapheresis session with single plasma exchange | Day 0, 1 hour after the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Genesia® after the plasmapheresis session with single plasma exchange | Day 0, 1 hour after the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the plasmapheresis session with single plasma exchange | Day 0, 4 hours after the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Genesia® after the plasmapheresis session with single plasma exchange | Day 0, 4 hours after the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels before the plasmapheresis session with single plasma exchange | Day 1
  Clauss functional method, g/L
Determination of fibrinogen levels with Genesia® before the plasmapheresis session with single plasma exchange | Day 1
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels before the plasmapheresis session with single plasma exchange | Day 3
  Clauss functional method, g/L
Determination of fibrinogen levels with Genesia® before the plasmapheresis session with single plasma exchange | Day 3
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the plasmapheresis session with single plasma exchange | Month 1, Day 1, 1 hour after the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Genesia® after the plasmapheresis session with single plasma exchange | Month 1, Day 1, 1 hour after the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the plasmapheresis session with single plasma exchange | Month 1, Day 4, 4 hours after the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Genesia® after the plasmapheresis session with single plasma exchange | Month 1, Day 4, 4 hours after the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the plasmapheresis session with single plasma exchange | Month 1, Day 3
  Clauss functional method, g/L
Determination of fibrinogen levels with Genesia® after the plasmapheresis session with single plasma exchange | Month 1, Day 3
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels before the first plasmapheresis session with double filtration plasmapheresis | Day 0, before the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® before the first plasmapheresis session with double filtration plasmapheresis | Day 0, before the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the first plasmapheresis session with double filtration plasmapheresis | Day 0, end of session
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® after the first plasmapheresis session with double filtration plasmapheresis | Day 0, end of session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the first plasmapheresis session with double filtration plasmapheresis | Day 0, 1 hour after the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® after the first plasmapheresis session with double filtration plasmapheresis | Day 0, 1 hour after the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the first plasmapheresis session with double filtration plasmapheresis | Day 0, 4 hours after the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® after the first plasmapheresis session with double filtration plasmapheresis | Day 0, 4 hours after the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels before the plasmapheresis session with double filtration plasmapheresis | Day 1
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® before the plasmapheresis session with double filtration plasmapheresis | Day 1
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels before the plasmapheresis session with double filtration plasmapheresis | Day 3
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® before the plasmapheresis session with double filtration plasmapheresis | Day 3
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the plasmapheresis session with double filtration plasmapheresis | Month 1, Day 1, 1 hour after the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® after the plasmapheresis session with double filtration plasmapheresis | Month 1, Day 1, 1 hour after the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the plasmapheresis session with double filtration plasmapheresis | Month 1, Day 1, 4 hours after the session
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® after the plasmapheresis session with double filtration plasmapheresis | Month 1, Day 1, 4 hours after the session
  Automated thrombin generation test on Génésia®.
Determination of fibrinogen levels after the plasmapheresis session with double filtration plasmapheresis | Month 1, Day 3
  Clauss functional method, g/L
Determination of fibrinogen levels with Génésia® after the plasmapheresis session with double filtration plasmapheresis | Month 1, Day 3
  Automated thrombin generation test on Génésia®.

SECONDARY OUTCOMES:
Complete blood count before the plasmapheresis session with single plasma exchange : White blood cells | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : White blood cells | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : White blood cells | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : White blood cells | Day 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : White blood cells | Day 3
  Quantitative, per microliter
Complete blood count before the plasmapheresis session with single plasma exchange : Red blood cells | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Red blood cells | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Red blood cells | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Red blood cells | Day 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Red blood cells | Day 3
  Quantitative, per microliter
Complete blood count before the plasmapheresis session with single plasma exchange : Hemoglobin | Day 0, Hour 0
  Quantitative, grams per liter
Complete blood count after the plasmapheresis session with single plasma exchange : Hemoglobin | Day 0, Hour 1
  Quantitative, grams per liter
Complete blood count after the plasmapheresis session with single plasma exchange : Hemoglobin | Day 0, Hour 4
  Quantitative, grams per liter
Complete blood count after the plasmapheresis session with single plasma exchange : Hemoglobin | Day 1
  Quantitative, grams per liter
Complete blood count after the plasmapheresis session with single plasma exchange : Hemoglobin | Day 3
  Quantitative, grams per liter
Complete blood count before the plasmapheresis session with single plasma exchange : Platelets | Day 0, Hour 0
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Platelets | Day 0, Hour 1
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Platelets | Day 0, Hour 4
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Platelets | Day 1
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Platelets | Day 3
  Quantitative, %
Complete blood count before the plasmapheresis session with single plasma exchange : Neutrophils | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Neutrophils | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Neutrophils | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Neutrophils | Day 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Neutrophils | Day 3
  Quantitative, per microliter
Complete blood count before the plasmapheresis session with single plasma exchange : Lymphocytes | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Lymphocytes | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Lymphocytes | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Lymphocytes | Day 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Lymphocytes | Day 3
  Quantitative, per microliter
Complete blood count before the plasmapheresis session with single plasma exchange : Monocytes | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Monocytes | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Monocytes | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Monocytes | Day 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Monocytes | Day 3
  Quantitative, per microliter
Complete blood count before the plasmapheresis session with single plasma exchange : Eosinophils | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Eosinophils | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Eosinophils | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Eosinophils | Day 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Eosinophils | Day 3
  Quantitative, per microliter
Complete blood count before the plasmapheresis session with single plasma exchange : Basophils | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Basophils | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Basophils | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Basophils | Day 1
  Quantitative, per microliter
Complete blood count after the plasmapheresis session with single plasma exchange : Basophils | Day 3
  Quantitative, per microliter
Complete blood count before the plasmapheresis session with single plasma exchange : Hematocrit | Day 0, Hour 0
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Hematocrit | Day 0, Hour 1
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Hematocrit | Day 0, Hour 4
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Hematocrit | Day 1
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Hematocrit | Day 3
  Quantitative, %
Complete blood count before the plasmapheresis session with single plasma exchange : Mean Corpuscular Volume | Day 0, Hour 0
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Volume | Day 0, Hour 1
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Volume | Day 0, Hour 4
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Volume | Day 1
  Quantitative, %
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Volume | Day 4
  Quantitative, %
Complete blood count before the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin | Day 0, Hour 0
  Quantitative, in pg
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin | Day 0, Hour 1
  Quantitative, in pg
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin | Day 0, Hour 4
  Quantitative, in pg
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin | Day 1
  Quantitative, in pg
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin | Day 3
  Quantitative, in pg
Complete blood count before the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin Concentration | Day 0, Hour 0
  Quantitative, in g/L
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin Concentration | Day 0, Hour 1
  Quantitative, in g/L
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin Concentration | Day 0, Hour 4
  Quantitative, in g/L
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin Concentration | Day 1
  Quantitative, in g/L
Complete blood count after the plasmapheresis session with single plasma exchange : Mean Corpuscular Hemoglobin Concentration | Day 3
  Quantitative, in g/L
Serum albumin before the plasmapheresis session with single plasma exchange | Day 0, Hour 0
  Quantitative, in g/dL
Serum albumin after the plasmapheresis session with single plasma exchange | Day 0, Hour 1
  Quantitative, in g/dL
Serum albumin after the plasmapheresis session with single plasma exchange | Day 0, Hour 4
  Quantitative, in g/dL
Serum albumin after the plasmapheresis session with single plasma exchange | Day 1
  Quantitative, in g/dL
Serum albumin after the plasmapheresis session with single plasma exchange | Day 3
  Quantitative, in g/dL
Prothrombin Time Test and International Normalized Ratio (PT/INR) before the plasmapheresis session with single plasma exchange | Day 0, Hour 0
  In seconds
Prothrombin Time Test and International Normalized Ratio (PT/INR) after the plasmapheresis session with single plasma exchange | Day 0, Hour 1
  In seconds
Prothrombin Time Test and International Normalized Ratio (PT/INR) after the plasmapheresis session with single plasma exchange | Day 0, Hour 4
  In seconds
Prothrombin Time Test and International Normalized Ratio (PT/INR) after the plasmapheresis session with single plasma exchange | Day 1
  In seconds
Prothrombin Time Test and International Normalized Ratio (PT/INR) after the plasmapheresis session with single plasma exchange | Day 3
  In seconds
Factors VIII, IX, XI and XII before the plasmapheresis session with single plasma exchange | Day 0, Hour 0
  By 1-stage APTT-based Factor assay, in seconds
Factors VIII, IX, XI and XII after the plasmapheresis session with single plasma exchange | Day 0, Hour 1
  By 1-stage APTT-based Factor assay, in seconds
Factors VIII, IX, XI and XII after the plasmapheresis session with single plasma exchange | Day 0, Hour 4
  By 1-stage APTT-based Factor assay, in seconds
Factors VIII, IX, XI and XII after the plasmapheresis session with single plasma exchange | Day 1
  By 1-stage APTT-based Factor assay, in seconds
Factors VIII, IX, XI and XII after the plasmapheresis session with single plasma exchange | Day 3
  By 1-stage APTT-based Factor assay, in seconds
Factors X, V and II [Prothrombin] before the plasmapheresis session with single plasma exchange | Day 0, Hour 0
  Prothrombin assay, in seconds
Factors X, V and II [Prothrombin] after the plasmapheresis session with single plasma exchange | Day 0, Hour 1
  Prothrombin assay, in seconds
Factors X, V and II [Prothrombin] after the plasmapheresis session with single plasma exchange | Day 0, Hour 4
  Prothrombin assay, in seconds
Factors X, V and II [Prothrombin] after the plasmapheresis session with single plasma exchange | Day 1
  Prothrombin assay, in seconds
Factors X, V and II [Prothrombin] after the plasmapheresis session with single plasma exchange | Day 3
  Prothrombin assay, in seconds
D-dimers and circulating soluble fibrin monomers before the plasmapheresis session with single plasma exchange | Day 0, Hour 0
  By enzyme-linked immunosorbent assay (ELISA) method
D-dimers and circulating soluble fibrin monomers after the plasmapheresis session with single plasma exchange | Day 0, Hour 1
  By enzyme-linked immunosorbent assay (ELISA) method
D-dimers and circulating soluble fibrin monomers after the plasmapheresis session with single plasma exchange | Day 0, Hour 4
  By enzyme-linked immunosorbent assay (ELISA) method
D-dimers and circulating soluble fibrin monomers after the plasmapheresis session with single plasma exchange | Day 1
  By enzyme-linked immunosorbent assay (ELISA) method
D-dimers and circulating soluble fibrin monomers after the plasmapheresis session with single plasma exchange | Day 3
  By enzyme-linked immunosorbent assay (ELISA) method
Platelet function test before the plasmapheresis session with single plasma exchange | Day 0, Hour 0
  ADP/collagen and adrenalin/collagen cartridges.
Platelet function test after the plasmapheresis session with single plasma exchange | Day 0, Hour 1
  ADP/collagen and adrenalin/collagen cartridges.
Platelet function test after the plasmapheresis session with single plasma exchange | Day 0, Hour 4
  ADP/collagen and adrenalin/collagen cartridges.
Platelet function test after the plasmapheresis session with single plasma exchange | Day 1
  ADP/collagen and adrenalin/collagen cartridges.
Platelet function test after the plasmapheresis session with single plasma exchange | Day 3
  ADP/collagen and adrenalin/collagen cartridges.
von Willebrand factor (vWF) activity - ristocetin cofactor test before the plasmapheresis session with single plasma exchange | Day 0, Hour 0
  Binding to platelet membrane glycoprotein Ib
von Willebrand factor (vWF) activity - ristocetin cofactor test after the plasmapheresis session with single plasma exchange | Day 0, Hour 1
  Binding to platelet membrane glycoprotein Ib
von Willebrand factor (vWF) activity - ristocetin cofactor test after the plasmapheresis session with single plasma exchange | Day 0, Hour 4
  Binding to platelet membrane glycoprotein Ib
von Willebrand factor (vWF) activity - ristocetin cofactor test after the plasmapheresis session with single plasma exchange | Day 1
  Binding to platelet membrane glycoprotein Ib
von Willebrand factor (vWF) activity - ristocetin cofactor test after the plasmapheresis session with single plasma exchange | Day 3
  Binding to platelet membrane glycoprotein Ib
Thrombin generation test on Génésia® before the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 0, Hour 0
  Triggered by 1 pM tissue factor
Thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 0, Hour 1
  Triggered by 1 pM tissue factor
Thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 0, Hour 4
  Triggered by 1 pM tissue factor
Thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 1
  Triggered by 1 pM tissue factor
Thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 3
  Triggered by 1 pM tissue factor
Automated thrombin generation test on Génésia® before the plasmapheresis session with single plasma exchange | Day 0, Hour 0
  Triggered by 5 pM tissue factor with response to purified thrombomodulin (thrombotic exploration version)
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange | Day 0, Hour 1
  Triggered by 5 pM tissue factor with response to purified thrombomodulin (thrombotic exploration version)
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange | Day 0, Hour 4
  Triggered by 5 pM tissue factor with response to purified thrombomodulin (thrombotic exploration version)
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange | Day 1
  Triggered by 5 pM tissue factor with response to purified thrombomodulin (thrombotic exploration version)
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange | Day 3
  Triggered by 5 pM tissue factor with response to purified thrombomodulin (thrombotic exploration version)
Complete blood count before the double filtration plasmapheresis session : White blood cells | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : White blood cells | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : White blood cells | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : White blood cells | Day 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : White blood cells | Day 3
  Quantitative, per microliter
Complete blood count before the double filtration plasmapheresis session : Red blood cells | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Red blood cells | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Red blood cells | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Red blood cells | Day 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Red blood cells | Day 4
  Quantitative, per microliter
Complete blood count before the double filtration plasmapheresis session : Hemoglobin | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Hemoglobin | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Hemoglobin | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Hemoglobin | Day 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Hemoglobin | Day 3
  Quantitative, per microliter
Complete blood count before the double filtration plasmapheresis session : Platelets | Day 0, Hour 0
  Quantitative, %
Complete blood count after the double filtration plasmapheresis session : Platelets | Day 0, Hour 1
  Quantitative, %
Complete blood count after the double filtration plasmapheresis session : Platelets | Day 0, Hour 4
  Quantitative, %
Complete blood count after the double filtration plasmapheresis session : Platelets | Day 1
  Quantitative, %
Complete blood count after the double filtration plasmapheresis session : Platelets | Day 3
  Quantitative, %
Complete blood count before the double filtration plasmapheresis session : Neutrophils | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Neutrophils | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Neutrophils | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Neutrophils | Day 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Neutrophils | Day 3
  Quantitative, per microliter
Complete blood count before the double filtration plasmapheresis session : Lymphocytes | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Lymphocytes | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Lymphocytes | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Lymphocytes | Day 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Lymphocytes | Day 3
  Quantitative, per microliter
Complete blood count before the double filtration plasmapheresis session : Monocytes | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Monocytes | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Monocytes | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Monocytes | Day 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Monocytes | Day 3
  Quantitative, per microliter
Complete blood count before the double filtration plasmapheresis session : Eosinophils | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Eosinophils | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Eosinophils | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Eosinophils | Day 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Eosinophils | Day 3
  Quantitative, per microliter
Complete blood count before the double filtration plasmapheresis session : Basophils | Day 0, Hour 0
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Basophils | Day 0, Hour 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Basophils | Day 0, Hour 4
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Basophils | Day 1
  Quantitative, per microliter
Complete blood count after the double filtration plasmapheresis session : Basophils | Day 3
  Quantitative, per microliter
Complete blood count before the double filtration plasmapheresis session : Hematocrit | Day 0, Hour 0
  Quantitative, %
Complete blood count after the double filtration plasmapheresis session : Hematocrit | Day 0, Hour 1
  Quantitative, %
Complete blood count after the double filtration plasmapheresis session : Hematocrit | Day 0, Hour 4
  Quantitative, %
Complete blood count after the double filtration plasmapheresis session : Hematocrit | Day 1
  Quantitative, %
Complete blood count after the double filtration plasmapheresis session : Hematocrit | Day 3
  Quantitative, %
Complete blood count before the double filtration plasmapheresis session : Mean Corpuscular Volume | Day 0, Hour 0
  Quantitative, fL
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Volume | Day 0, Hour 1
  Quantitative, fL
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Volume | Day 0, Hour 4
  Quantitative, fL
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Volume | Day 1
  Quantitative, fL
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Volume | Day 3
  Quantitative, fL
Complete blood count before the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin | Day 0, Hour 0
  Quantitative, pg
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin | Day 0, Hour 1
  Quantitative, pg
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin | Day 0, Hour 4
  Quantitative, pg
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin | Day 1
  Quantitative, pg
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin | Day 3
  Quantitative, pg
Complete blood count before the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin Concentration | Day 0, Hour 0
  Quantitative, g/L
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin Concentration | Day 0, Hour 1
  Quantitative, g/L
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin Concentration | Day 0, Hour 4
  Quantitative, g/L
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin Concentration | Day 1
  Quantitative, g/L
Complete blood count after the double filtration plasmapheresis session : Mean Corpuscular Hemoglobin Concentration | Day 3
  Quantitative, g/L
Serum albumin before the double filtration plasmapheresis session. | Day 0, Hour 0
  Quantitative, g/L
Serum albumin after the double filtration plasmapheresis session. | Day 0, Hour 1
  Quantitative, g/L
Serum albumin after the double filtration plasmapheresis session. | Day 0, Hour 4
  Quantitative, g/L
Serum albumin after the double filtration plasmapheresis session. | Day 1
  Quantitative, g/L
Serum albumin after the double filtration plasmapheresis session. | Day 3
  Quantitative, g/L
Prothrombin Time Test and International Normalized Ratio (PT/INR) before the double filtration plasmapheresis session. | Day 0, Hour 0
  In seconds
Prothrombin Time Test and International Normalized Ratio (PT/INR) after the double filtration plasmapheresis session. | Day 0, Hour 1
  In seconds
Prothrombin Time Test and International Normalized Ratio (PT/INR) after the double filtration plasmapheresis session. | Day 0, Hour 4
  In seconds
Prothrombin Time Test and International Normalized Ratio (PT/INR) after the double filtration plasmapheresis session. | Day 1
  In seconds
Prothrombin Time Test and International Normalized Ratio (PT/INR) after the double filtration plasmapheresis session. | Day 3
  In seconds
Factors VIII, IX, XI and XII before the double filtration plasmapheresis session. | Day 0, Hour 0
  1-stage APTT-based Factor assay
Factors VIII, IX, XI and XII after the double filtration plasmapheresis session. | Day 0, Hour 1
  1-stage APTT-based Factor assay
Factors VIII, IX, XI and XII after the double filtration plasmapheresis session. | Day 0, Hour 4
  1-stage APTT-based Factor assay
Factors VIII, IX, XI and XII after the double filtration plasmapheresis session. | Day 1
  1-stage APTT-based Factor assay
Factors VIII, IX, XI and XII after the double filtration plasmapheresis session. | Day 3
  1-stage APTT-based Factor assay
Factors X, V and II [Prothrombin] before the double filtration plasmapheresis session. | Day 0, Hour 0
  Prothrombin assay, in seconds
Factors X, V and II [Prothrombin] after the double filtration plasmapheresis session. | Day 0, Hour 1
  Prothrombin assay, in seconds
Factors X, V and II [Prothrombin] after the double filtration plasmapheresis session. | Day 0, Hour 4
  Prothrombin assay, in seconds
Factors X, V and II [Prothrombin] after the double filtration plasmapheresis session. | Day 1
  Prothrombin assay, in seconds
Factors X, V and II [Prothrombin] after the double filtration plasmapheresis session. | Day 3
  Prothrombin assay, in seconds
D-dimers and circulating soluble fibrin monomers before the double filtration plasmapheresis session. | Day 0, Hour 0
  By enzyme-linked immunosorbent assay (ELISA) method
D-dimers and circulating soluble fibrin monomers after the double filtration plasmapheresis session. | Day 0, Hour 1
  By enzyme-linked immunosorbent assay (ELISA) method
D-dimers and circulating soluble fibrin monomers after the double filtration plasmapheresis session. | Day 0, Hour 4
  By enzyme-linked immunosorbent assay (ELISA) method
D-dimers and circulating soluble fibrin monomers after the double filtration plasmapheresis session. | Day 1
  By enzyme-linked immunosorbent assay (ELISA) method
D-dimers and circulating soluble fibrin monomers after the double filtration plasmapheresis session. | Day 3
  By enzyme-linked immunosorbent assay (ELISA) method
Platelet function test before the double filtration plasmapheresis session. | Day 0, Hour 0
  ADP/collagen and adrenalin/collagen cartridges
Platelet function test after the double filtration plasmapheresis session. | Day 0, Hour 1
  ADP/collagen and adrenalin/collagen cartridges
Platelet function test after the double filtration plasmapheresis session. | Day 0, Hour 4
  ADP/collagen and adrenalin/collagen cartridges
Platelet function test after the double filtration plasmapheresis session. | Day 1
  ADP/collagen and adrenalin/collagen cartridges
Platelet function test after the double filtration plasmapheresis session. | Day 3
  ADP/collagen and adrenalin/collagen cartridges
von Willebrand factor (vWF) activity - ristocetin cofactor test before the double filtration plasmapheresis session. | Day 0, Hour 0
  Binding to platelet membrane glycoprotein Ib
von Willebrand factor (vWF) activity - ristocetin cofactor test after the double filtration plasmapheresis session. | Day 0, Hour 1
  Binding to platelet membrane glycoprotein Ib
von Willebrand factor (vWF) activity - ristocetin cofactor test after the double filtration plasmapheresis session. | Day 0, Hour 4
  Binding to platelet membrane glycoprotein Ib
von Willebrand factor (vWF) activity - ristocetin cofactor test after the double filtration plasmapheresis session. | Day 1
  Binding to platelet membrane glycoprotein Ib
von Willebrand factor (vWF) activity - ristocetin cofactor test after the double filtration plasmapheresis session. | Day 3
  Binding to platelet membrane glycoprotein Ib
Automated thrombin generation test on Génésia® before the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 0, Hour 0
  Triggered by 1 pM tissue factor
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 0, Hour 1
  Triggered by 1 pM tissue factor
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 0, Hour 4
  Triggered by 1 pM tissue factor
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 1
  Triggered by 1 pM tissue factor
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (hemorrhagic exploration version) | Day 3
  Triggered by 1 pM tissue factor
Automated thrombin generation test on Génésia® before the plasmapheresis session with single plasma exchange (thrombotic exploration version) | Day 0, Hour 0
  Triggered by 5 pM tissue factor with response to purified thrombomodulin
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (thrombotic exploration version) | Day 0, Hour 1
  Triggered by 5 pM tissue factor with response to purified thrombomodulin
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (thrombotic exploration version) | Day 0, Hour 4
  Triggered by 5 pM tissue factor with response to purified thrombomodulin
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (thrombotic exploration version) | Day 1
  Triggered by 5 pM tissue factor with response to purified thrombomodulin
Automated thrombin generation test on Génésia® after the plasmapheresis session with single plasma exchange (thrombotic exploration version) | Day 3
  Triggered by 5 pM tissue factor with response to purified thrombomodulin
Plasma Bank | Before Day 0, hour 0
  Storage of unused tube ends
Plasma Bank | Day 0, hour1
  Storage of unused tube ends
Plasma Bank | Day 0, hour 4
  Storage of unused tube ends
Plasma Bank | Day 1
  Storage of unused tube ends
Plasma Bank | Day 3
  Storage of unused tube ends
Plasma Bank | After end of session Day 0, H0
  Storage of unused tube ends

OTHER OUTCOMES:
Gender of patients | Day 0, Hour 0
  Recorded as Male, Female, Nonbinary
Age of patients | Day 0, Hour 0
  Recorded in years
Weight of patients | Day 0, Hour 0
  Recorded in kilos
Height of patients | Day 0, Hour 0
  Recorded in centimeters
Diagnostic history of patients | Day 0, Hour 0
  The patients' diagnostic history will be recorded
Patient's apheresis protocol | Day 0, Hour 0
  The apheresis protocol used, and parameters related to plasmapheresis will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Emilie PAMBRUN, Docteur, Principal Investigator — Nîmes University Hospital; Sylvie BOUVIER, Docteur, Principal Investigator — Nîmes University Hospital; Jean-Christophe GRIS, Professor, Principal Investigator — Nîmes University Hospital; Mathieu FORTIER, Principal Investigator — Nîmes University Hospital
Locations (1):
- CHU de Nîmes, Nîmes, France